CLINICAL TRIAL: NCT00004278
Title: Phase III Randomized, Controlled Study of Ganciclovir for Symptomatic Congenital Cytomegalovirus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/11689; NIAID-558607
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-07

CONDITIONS: Cytomegalovirus Infections
Keywords: congenital cytomegalovirus infection; cytomegalovirus infection; herpesvirus infection; immunologic disorders and infectious disorders; neonatal disorders; rare disease; viral infection
MeSH Terms: conditions — Cytomegalovirus Infections; Herpesviridae Infections; Immune System Diseases; Communicable Diseases; Infant, Newborn, Diseases; Rare Diseases; Virus Diseases | interventions — Ganciclovir

INTERVENTIONS:
Drug: ganciclovir

SUMMARY:
OBJECTIVES:

I. Evaluate the efficacy of ganciclovir (12 mg/kg per day) versus no treatment in neonates with symptomatic congenital cytomegalovirus infection with central nervous system disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Patients are stratified by participating institution.

Patients are randomly assigned to no antiviral therapy or intravenous ganciclovir every 12 hours for 6 weeks.

Patients are followed at weeks 1-4 and 12, months 6, 12, 24, 36, 48, and 60, and yearly thereafter until puberty (when possible).

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Symptomatic cytomegalovirus (CMV) infection: Central nervous system disease, with or without other organ system involvement, e.g.: Microcephaly, i.e., less than 5% for age Radiologic changes indicating brain disease Cerebrospinal fluid exam abnormal for age Chorioretinitis Hearing defects
* CMV confirmed by urine, throat, buffy coat, and/or conjunctiva culture
* No hydroencephalopathy or other devastating brain involvement

--Prior/Concurrent Therapy--

* No concurrent antiviral agent No concurrent immune globulin

--Patient Characteristics--

* Age: Under 1 month (preferably under 2 weeks)
* Life expectancy: No imminent demise
* Renal: Creatinine no greater than 1.5 mg/dL
* Other: Birth weight at least 1200 g Gestational age at least 32 weeks No HIV infection No concurrent bacterial infection Eligible if resolved following 2-week treatment and CMV symptoms persist

Ages: 0 Years to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130
Dates: Start 1991-12

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Whitley, Study Chair